CLINICAL TRIAL: NCT01966679
Title: Targeting GABA-A for the Treatment of Social Disability in Young Adults With Autism Spectrum Disorders: A Phase II Proof of Mechanism Trial
Acronym: FAST-AS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, James McCracken, Department Chair, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHS-NIH-DA-12-241
Record Dates: First submitted 2013-10-08; First posted 2013-10-21 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double-blind (active versus placebo) (Active Comparator): AZD7325 versus placebo
  Interventions: Drug: AZD7325
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7325
  Other Names: sugar pill
  Arms: Double-blind (active versus placebo)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is a NIMH-funded multi-site clinical trial that includes UCLA as the coordinating site, with Emory University and Seattle Children's Hospital, as other recruiting sites, and the Nathan Kline Institute as the Data Management Center. The purpose of the study is to examine the effects of an investigational drug, AZD7325, as a potential treatment for high-functioning adults 18 -35 years old with Autism Spectrum Disorders (ASD). The primary study measures are effects on brain waves as measured by non-invasive brain wave recordings (electroencephalograms or EEGs), assessments of side effects, and measures of attention and learning.

The study drug, AZD7325, is manufactured by Astra Zeneca, and was initially tested as a medication for anxiety disorders in over 488 subjects, but was not pursued for marketing due to too few benefits for anxiety. AZD7325 was found to have a very good safety profile and was tolerated by the majority of subjects. AZD7325 has some similar actions to currently marketed anxiety drugs in the benzodiazepine class, but lacks the sedative and negative effects on attention of the benzodiazepines. The study drug is designed to target the GABA neurotransmitter system which is believed to be abnormal in this population.

There are 2 study phases. Phase 1 includes the recruitment of 24 healthy volunteers without mental disorder (6 per site) in order to establish normal EEG reference ranges. Controls will only be seen for one study visit which includes a clinical evaluation, physical exam, routine blood tests, and an EEG. Once control recruitment is complete, Phase 2 will begin.

Phase 2 involves the recruitment of 40 adults (10 per site) 18 - 35 years old with a diagnosis of ASD, normal intelligence, and specific EEG patterns compared to control values. Screening for eligibility will be performed in one visit, which includes a clinical evaluation, tests of learning and intelligence, blood and urine tests, and an EEG. Those subjects who are found to be eligible will be enrolled in a 6-week medication study. Subjects with ASD who are enrolled will be randomly assigned to receive the study drug AZD7325 or placebo in matching capsules. Subjects will be seen weekly by study physicians and clincians for the 7 study visits, including 3 additional EEG recordings, and then for a final follow-up visit (9 total visits including screening lasting up to 11 weeks to complete). Study physicians can adjust the dose of study medication to reduce any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of ASD as defined by DSM-5, confirmed by clinical evaluation and supported by the Autism Diagnostic Observation Schedule (ADOS)
* Ages 18- 35 years inclusive
* IQ estimate of >80
* Aberrant Behavior Checklist (ABC)-Social Withdrawal Score >10 (>40% over population mean for developmentally disabled adults)
* Existing allowed concomitant medication treatment stable for the 8 weeks prior to study entry, and no anticipated changes
* Ability to comply with all protocol procedures and assessments
* Availability of a reliable parent or caregiver willing to provide information regarding subject behavior and health status
* Evidence of EEG biomarker deficit as defined below.

Exclusion Criteria:

* Evidence of current drug or alcohol abuse or dependence
* Prior history of drug or alcohol abuse or dependence in prior 12 months
* History of seizure disorder (except febrile seizures)
* Clinically significant aggressive, disruptive, or suicidal behavior in the 3 months prior to study enrollment
* Presence of a chronic medical condition or prohibited medication (see list in Human Subjects section) which would potentially interfere with the assessment of treatment effects, or interact with study medications (eg. hepatic, neurologic, renal disease) to increase risk to the subject
* History of paradoxical reactions to benzodiazepines
* Clinically significant deviation from the reference range in clinical laboratory test results at screening, as judged by the investigator
* ALT or AST greater than the upper limit of the laboratory standard reference range at screening
* EKG abnormalities considered to be clinically significant as determined by the investigator and confirmed by an experienced cardiologist
* Fredericia-corrected QT (QTcF) interval of >450 msec
* Clinical judgment of the study physician of inability to perform the requirements of the study
* For sexually active female and male subjects, refusal to agree to maintain a double-barrier birth control method during protocol participation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
EEG | week 6

CONTACTS AND LOCATIONS:
Overall Officials: James McCracken, MD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - UCLA, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Seattle Children's Research Institute, Seattle, Washington

REFERENCES:
- See also: Related Info — http://autism.ucla.edu